CLINICAL TRIAL: NCT06162403
Title: Exploring the Benefit of Peripheral Nerve Stimulation in Treating Pain From Chemo-induced Peripheral Neuropathy: A Longitudinal Single Center Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0368; NCI-2023-10303 (Other: NCI-2023-10303)
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Nerve Stimulation; Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peripheral Nerve Stimulation (Experimental): Participants will be asked to have PNS leads inserted via a needle, which will provide a mild, stimulating electrical current to the effected nerves 24 hours a day for up to 60 days. Participants will have study visits during and after this time.
  Interventions: Other: Peripheral Nerve Stimulation

INTERVENTIONS:
Other: Peripheral Nerve Stimulation — The leads are inserted through a needle. If needed, the study team may give participants anesthetic (for example, as a cream/gel on your skin and/or as an injection) to numb the area where the leads will be injected.

SUMMARY:
To learn if peripheral nerve stimulation (PNS) can help to improve pain in participants with CIPN.

DETAILED DESCRIPTION:
Primary objective:

To assess Pain intensity (NRS) scores in chemotherapy induced peripheral neuropathy (CIPN) participants before and after use of peripheral nerve stimulation (PNS).

Secondary objectives:

To assess changes in quantitative sensory testing (QST), gait testing, and skin punch biopsy to compare the integrity of Meissner's corpuscles (MC), pain disability using the Oswestry Disability Index (ODI), pain interference using the Brief Pain Inventory (BPI), and Patient Global Impression of Change (PGIC) in CIPN patients before and after use of PNS.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with chronic (≥90 days duration) CIPN (due to either vinca alkaloids, taxanes, bortezomib, thalidomide, platinum-based compounds or ionizing irradiation) of the lower extremity, seen at Pain Management Center at MD Anderson Cancer Center
* Participants reports baseline pain ≥ 4 (0-10 scale, NRS)
* Participants between ages 18-85 years old
* Participants who have completed chemotherapy within the previous year at the time of enrollment

Exclusion Criteria:

* Participants with cognitive dysfunction
* Participants with recent history (<6 months) of drug or alcohol abuse
* Participants with open skin lesion or undergoing antibiotic therapy for local for systemic infection
* Participants with allergies to local anesthesia, steroids, or adhesives
* Participants with conditions that conflict with the SPRINT PNS System Indications for Use, including Contraindications and Warnings.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Saba Javed, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org